CLINICAL TRIAL: NCT04924205
Title: A Prospective Comparison Of Primary Total Knee Arthroplasty Rehabilitation Using A Smart Orthotic Versus Outpatient Physical Therapy
Brief Title: A Comparison Of Primary TKA Rehabilitation Using A Smart Orthotic Versus Outpatient Physical Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolas Noiseux, MD, MS, FRCSC (Other)
Responsible Party: Sponsor-Investigator, Nicolas Noiseux, MD, MS, FRCSC, Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202002141
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Arthropathy of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient Physical Therapy (No Intervention)
- Smart Orthotic Device (FM2 Knee Brace) (Experimental)
  Interventions: Device: FM2 Knee Brace

INTERVENTIONS:
Device: FM2 Knee Brace — Participants in this group will use the FM2 Knee Brace for their post-TKA physical therapy.
  Arms: Smart Orthotic Device (FM2 Knee Brace)

SUMMARY:
This will be a prospective, randomized, noninferiority clinical trial comparing rehabilitation methods post-total knee arthroplasty (TKA). Population of interest is adult hip/knee clinic patients over age 18 who are indicated for unilateral primary total knee arthroplasty. All TKA patients are prescribed physical therapy (PT) for rehabilitation post-operatively. The investigators will compare this current treatment with a new, validated, wearable smart knee brace (FM2 Knee Brace) that can be used for rehabilitation post-TKA. Following enrollment in the study, the investigators will match and randomize participants into two cohorts (outpatient PT versus FM2 Knee Brace). Outpatient PT group will be prescribed routine six-week course of outpatient PT (no pool exercises, remainder at therapist's discretion) to start as soon as possible upon discharge. The FM2 Knee Brace group will complete device set up at pre-op visit and will be prescribed 3-4 exercises to complete at their discretion over six weeks. The investigators will collect measurements of knee flexion, extension, total arc of motion at pre-op visit and at 6-week, 3-month, and 1-year post-op visits. The investigators will also plan to record additional PROs, therapy compliance, and complication rates. The investigators will compare the two groups to test whether the new FM2 Knee Brace is noninferior to regular PT when recovering from TKA, and if the new technology could be an alternative to outpatient PT.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-100
* Indicated for primary total knee arthroplasty
* Possess a smartphone with capabilities to use the FocusMotion app and FM2 Knee Brace
* Home discharge post-operatively

Exclusion Criteria:

* Prior ipsilateral knee surgery
* Prior manipulation under anesthesia of either knee
* BMI > 40

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | pre-surgery
  The study will collect measurements of knee flexion, extension, total arc of motion, and will also plan to record therapy compliance and complication rates. The two groups will be compared to study if the FM2 Knee Brace group is clinically non-inferior to the standard PT group with respect to knee range of motion.
Range of Motion | 6 weeks post-surgery
  The study will collect measurements of knee flexion, extension, total arc of motion, and will also plan to record therapy compliance and complication rates. The two groups will be compared to study if the FM2 Knee Brace group is clinically non-inferior to the standard PT group with respect to knee range of motion.
Range of Motion | 3 months post-surgery
  The study will collect measurements of knee flexion, extension, total arc of motion, and will also plan to record therapy compliance and complication rates. The two groups will be compared to study if the FM2 Knee Brace group is clinically non-inferior to the standard PT group with respect to knee range of motion.
Range of Motion | 1 year post-surgery
  The study will collect measurements of knee flexion, extension, total arc of motion, and will also plan to record therapy compliance and complication rates. The two groups will be compared to study if the FM2 Knee Brace group is clinically non-inferior to the standard PT group with respect to knee range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No